CLINICAL TRIAL: NCT06538259
Title: Effects of Transcranial Direct Current Stimulation Combined With Retrieval Practice on Semantic Memory in Patients With Schizophrenia
Brief Title: Effects of tDCS Combined With Retrieval Practice on Semantic Memory in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeast Normal University (Other)
Responsible Party: Principal Investigator, Xiaofeng Ma, Professor, Northeast Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No.2023023
Record Dates: First submitted 2024-07-27; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Schizophrenic Patients
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anodal group (Experimental): In the anodal group, the anode was placed over the left DLPFC (F3), and the cathode was placed over the contralateral supraorbital area (FP2). A direct current of 2mA was applied for 20 minutes during each stimulation session. Stimulation was conducted twice a day, at 9 a.m. and 2 p.m., for 5 consecutive days, totaling 10 sessions.
  Interventions: Device: Transcranial direct current stimulation (tDCS)-anodal group
- sham group (Sham Comparator): In the sham group, the stimulation parameters, including the stimulation site and duration, were identical to those of the anodal group. However, during the 10-second ramp-up and ramp-down periods before and after stimulation, patients were unaware that the current was turned off.
  Interventions: Device: Transcranial direct current stimulation (tDCS)-sham group

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS)-anodal group — 2mA/20mins/session; 2sessions/day,5days
  Arms: anodal group
Device: Transcranial direct current stimulation (tDCS)-sham group — 0mA/20mins/session; 2sessions/day,5days
  Arms: sham group

SUMMARY:
The semantic processing deficit stands as a central feature of cognitive abnormalities in schizophrenia. Both transcranial direct current stimulation (tDCS) and retrieval practice have been demonstrated as external techniques capable of ameliorating the semantic processing deficit in individuals with schizophrenia. The inquiry examines whether the combined effect of tDCS and retrieval practice, following tDCS intervention targeting the left dorsolateral prefrontal cortex (L-DLPFC) in patients with schizophrenia, contributes to the preservation of semantic memory in these individuals.

Investigators recruited 52 patients diagnosed with schizophrenia from hospitals. After five consecutive days of tDCS intervention (2 mA × 20 mins, twice per day), Investigators administered a word list memorization task comparing retrieval practice and restudy strategies. Subsequently, Investigators observed their immediate and delayed memory performance through tests.

DETAILED DESCRIPTION:
Treatment was administered by two examiners, and after a total of 10 sessions over 5 consecutive days, a final group of 52 patients participated in the learning and testing phase. Among them, 27 received anodal stimulation, while 25 received sham stimulation. Each participant of each stimulation type was involved in both learning conditions, meaning that all participants completed both retrieval and restudy learning and testing.

1. Stimulation phase:

   In the anodal group, the anode was placed over the left DLPFC (F3), and the cathode was placed over the contralateral supraorbital area (FP2). A direct current of 2mA was applied for 20 minutes during each stimulation session. Stimulation was conducted twice a day, at 9 a.m. and 2 p.m., for 5 consecutive days, totaling 10 sessions. In the sham group, the stimulation parameters, including the stimulation site and duration, were identical to those of the anodal group. However, during the 10-second ramp-up and ramp-down periods before and after stimulation, patients were unaware that the current was turned off.
2. Learning phase:

   The experimental procedure followed the classic retrieval practice paradigm, which included a learning phase and a final test phase.

   During the experiment, participants were informed that they would learn two lists of words. Subsequently, they might either learn the words again or complete a list recall test, and will be given a final test shortly thereafter. The learning of the retrieval practice list and the restudy list was conducted in a randomly balanced manner. Each word was presented for 5 seconds, with a 500-millisecond interval between words. To avoid providing secondary retrieval cues between examples, all words were shuffled pseudo-randomly within categories. Each list contained 17 words, consisting of 5 examples from each of the 3 experimental categories (15 experimental examples, 2 filler examples). The first and last words presented in each list were filler words, thus controlling for the primacy and recency effects on memory.

   For the retrieval practice list, participants underwent two learning sessions and two retrieval sessions (S-T-S-T). During retrieval, participants were instructed to write down all the words they had just remembered within 5 minutes. For the restudy list, participants underwent four study sessions (S-S-S-S). Between each learning cycle, participants completed a 3-minute simple arithmetic task (dispersed attention task).
3. Testing phase:

Immediate Test: Participants were instructed to recall as many words as possible from the learned lists within 10 minutes after completing all learning tasks.

Delayed Test: Participants were informed to recall as many words as possible from the learned lists within 10 minutes 24 hours later.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the diagnostic criteria for schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5);
2. Aged 18 years or older, regardless of gender, with an educational level of elementary school or above;
3. All patients received stable-level antipsychotic medication treatment, were in a stable phase of disease treatment, able to understand the testing requirements, and cooperated to complete all research tasks;
4. No history of neurological disorders or other serious physical illnesses, and no history of intellectual disability;
5. No color blindness, color weakness, or other color vision impairments, with normal vision or corrected vision.

Exclusion Criteria:

1. Clear cognitive impairment caused by somatic or cerebral organic lesions, such as cerebrovascular diseases, traumatic brain injury, etc;
2. Individuals with mental disorders caused by substance dependence or abuse, or the use of psychoactive substances;
3. History of brain injury or other central nervous system-related organic diseases;
4. Individuals at significant risk of suicide or harming others;
5. Participation in similar experiments in the past 30 days prior to baseline.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
The correct recall rate of word lists | 5mins to 24 hours
  The correct recall rate of word lists was calculated for each subject by the experimental assistant.
Adjusted Ratio of Clustering (ARC) | 5mins to 24 hours
  Free recall organization was measured by the Adjusted Ratio of Clustering (ARC) scores

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Ma, Professor, Principal Investigator — Northwest Normal University
Locations (1):
- Northwest Normal University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavendish BA, de Lima MFR, Pericoli L, Buratto LG. Effects of combining retrieval practice and tDCS over long-term memory: A randomized controlled trial. Brain Cogn. 2022 Feb;156:105807. doi: 10.1016/j.bandc.2021.105807. Epub 2021 Dec 20. PMID 34949566
- [Background] Javadi AH, Walsh V. Transcranial direct current stimulation (tDCS) of the left dorsolateral prefrontal cortex modulates declarative memory. Brain Stimul. 2012 Jul;5(3):231-241. doi: 10.1016/j.brs.2011.06.007. Epub 2011 Jul 26. PMID 21840287
- [Background] Sreeraj VS, Bose A, Chhabra H, Shivakumar V, Agarwal SM, Narayanaswamy JC, Rao NP, Kesavan M, Varambally S, Venkatasubramanian G. Working memory performance with online-tDCS in schizophrenia: A randomized, double-blinded, sham-controlled, partial cross-over proof-of-concept study. Asian J Psychiatr. 2020 Apr;50:101946. doi: 10.1016/j.ajp.2020.101946. Epub 2020 Feb 11. PMID 32087502
- [Background] Guimond S, Hawco C, Lepage M. Prefrontal activity and impaired memory encoding strategies in schizophrenia. J Psychiatr Res. 2017 Aug;91:64-73. doi: 10.1016/j.jpsychires.2017.02.024. Epub 2017 Mar 8. PMID 28325680
- [Background] Kim J, Iwata Y, Plitman E, Caravaggio F, Chung JK, Shah P, Blumberger DM, Pollock BG, Remington G, Graff-Guerrero A, Gerretsen P. A meta-analysis of transcranial direct current stimulation for schizophrenia: "Is more better?". J Psychiatr Res. 2019 Mar;110:117-126. doi: 10.1016/j.jpsychires.2018.12.009. Epub 2018 Dec 10. PMID 30639917
- [Background] Jantzi C, Mengin AC, Serfaty D, Bacon E, Elowe J, Severac F, Meyer N, Berna F, Vidailhet P. Retrieval practice improves memory in patients with schizophrenia: new perspectives for cognitive remediation. BMC Psychiatry. 2019 Nov 11;19(1):355. doi: 10.1186/s12888-019-2341-y. PMID 31711448
- [Derived] Pan W, Li T, Ma X, Huo X. Effects of transcranial direct current stimulation combined with retrieval practice on semantic memory in patients with schizophrenia. BMC Psychiatry. 2025 Mar 7;25(1):214. doi: 10.1186/s12888-025-06530-y. PMID 40055696

DOCUMENTS (2):
  • Study Protocol (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT06538259/Prot_000.pdf
  • Informed Consent Form (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT06538259/ICF_001.pdf